CLINICAL TRIAL: NCT00381914
Title: Vitamin D Dose-Response Study to Establish Dietary Requirements in Infants
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: McGill University (Other)
Responsible Party: Principal Investigator, Hope Weiler, Associate Professor, McGill University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: HW-06-01
Record Dates: First submitted 2006-09-27; First posted 2006-09-28 (Estimated); Last update posted 2012-03-02 (Estimated); Status verified 2012-03

CONDITIONS: Vitamin D Deficiency
Keywords: Infants; Vitamin D; Dose-response
MeSH Terms: conditions — Vitamin D Deficiency | interventions — Vitamin D

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 (Experimental): 400 IU / day vitamin D
  Interventions: Drug: Vitamin D
- 2 (Experimental): 800 IU / day vitamin D
  Interventions: Drug: Vitamin D
- 3 (Experimental): 1200 IU / day vitamin D
  Interventions: Drug: Vitamin D

INTERVENTIONS:
Drug: Vitamin D — 400 IU vitamin D / day
  Arms: 1
Drug: Vitamin D — 800 IU vitamin D / day
  Arms: 2
Drug: Vitamin D — 1200 IU vitamin D / day
  Arms: 3

SUMMARY:
The research team is comprised of an expert nutrition scientist and a pediatrician with expertise in endocrinology. Both have world-class experience in assessing bone mass in infancy. Together they have designed a study to determine how much dietary vitamin D is needed to optimize health in infants. This is important since many infants are born with vitamin D deficiency. At present the dosage of vitamin D that is optimal for infant health is unclear and recent research suggests that vitamin D status very early in life has long lasting effects on bone mass and other health issues. Therefore, in a group of healthy infants, this research team will test which dosage of vitamin D is needed to achieve optimal vitamin D status. Optimal vitamin D status will be based on growth, biomarkers of vitamin D and bone status in blood and also general health. The infants will all be breastfed and begin the study at about 2 weeks of age. At 3 months intervals over the first year of life, each infant will be measured for growth, duration of breastfeeding and supplement use plus have a bone density scan to determine changes in bone growth. The data will be helpful to guide health care professionals in providing the best care possible for their infants. It will also be important to the health of populations since dietary recommendations for vitamin D are used to guide fortification of foods and development of evidence based policy around nutrient recommendations and their implementation.

DETAILED DESCRIPTION:
Vitamin D status is currently judged by serum 25(OH)D and the parathyroid hormone (PTH)-25(OH)D dynamic (1). The ultimate effect of vitamin D on human health is a healthy skeleton, which is characterized in infancy by normal linear growth and bone mineral accretion and absence of bone related disease, such as rickets (1). The importance of these indicators is illustrated in epidemiological research, where linear growth in infancy is positively related to peak bone mass as an adult (2). Moreover, both vitamin D status (3) and intake (4) in infancy are related to bone mass in children.

In 2004, Health Canada reaffirmed its population health policy that all breastfed, healthy term infants in Canada receive a daily vitamin D3 supplement of 400 IU (5). This policy recommendation was made in consultation with the Canadian Expert Advisory Committee on Dietary Reference Intakes (DRI). They determined that the 1997 DRI value for vitamin D of 200 IU was too low for Canadians based on Canadian studies (6, 7) and surveillance systems (1) that indicated a high rate of vitamin D deficiency and vitamin D deficient rickets continued in Canada.

Both the Health Canada committee (5) and Institute of Medicine Committee on Dietary Recommended Intakes (1) acknowledged that there was considerable uncertainty regarding what defines optimal vitamin D intake in infancy based on functional outcomes.

In adults, a minimum serum 25(OH)D value of 75 nmol/L now defines optimal vitamin D status (8). This concentration is derived from dose-response studies of the relationship between 25(OH)D and PTH, where PTH plateaus in approximately the mid-normal range and also from studies where 25(OH)D concentrations between 90 and 100 nmol/L are positively related to bone mineral density (BMD) in young adults (9). A dose-response study to determine the physiological and functional response to vitamin D3 supplementation has not been conducted in infants and is necessary to confidently set DRI values for Canadian infants.

In summary, health care professionals are faced with major gaps in knowledge of: a) what constitutes optimal vitamin D status in infancy based on the physiological and functional outcomes, 25(OH)D, PTH and bone mass; and b) what oral dosage of vitamin D supplement is required to elevate serum 25(OH)D to optimal values as the key biomarker of optimal vitamin D status.

The global objective of this study is to conduct a dose-response study of vitamin D3 intakes and to provide information regarding the physiological and functional response to vitamin D supplementation in infancy, including: 25(OH)D concentrations and the relationship between 25(OH)D, PTH and bone mineral accretion. Once the best dosage is determined, funding for a larger study spanning all Canadian regions will be sought to more conclusively demonstrate that this dosage is appropriate for all Canadian infants. In the larger study, infants will be followed longitudinally to confirm that optimization of vitamin D status in infancy enhances peak bone mass.

2.0 BACKGROUND 2.1 Recommendations for Intakes of Vitamin D for Infants The AI value of at least 200 IU/d was derived from the amount of breast milk typically consumed by infants and the concentration of vitamin D in breast milk that resulted in serum 25(OH)D concentrations above 27.5 nmol/L (1). The current recommendations for vitamin D intake in Canada for infants are listed below, but no dosage has been evaluated using dose-response studies conducted in Canada.

* 400 IU vitamin D3/d for infants recommended in 2004 by Health Canada, The Canadian Pediatric Society and Dietitians of Canada in Guidelines for Healthy Term Infants (5); and
* that entirely breast-fed infants should be given 400 IU of vitamin D daily that may be increased to 800 IU/d from October through April as recommended by the Indian and Inuit Committee of the Canadian Pediatric Society (10). Infants bottle-fed formulas made from fortified whole or canned milk should receive additional 400 IU from October through April (10).

2.2 Vitamin D Metabolism and Sources of Vitamin D for Infants: The Canadian Scenario Endogenously synthesized vitamin D is in the form of cholecalciferol (vitamin D3). Most food sources and supplements in Canada have this mammalian form, but some contain the plant form, ergocalciferol (vitamin D2). Vitamin D3 is estimated to be approximately 9.5 times more potent than vitamin D2 (12).

Endogenous synthesis accounts for the majority of vitamin D in adults (8). Above latitude 42 in the northern hemisphere, synthesis is limited to late spring through mid-autumn, because of the low intensity of UVB radiation, during the rest of the year. The majority of Canadians reside north of the 42nd parallel, placing them at risk for hypovitaminosis D year round because of the use of sunscreen and environmental factors, such as clothing and pollution, which reduce exposure to UVB sunlight (14). This means that endogenous synthesis in pregnant women and subsequent maternal-fetal transfer may be compromised. Fortified foods such as milk, margarine and vitamin supplements remain the major source of vitamin D for many Canadian adults.

2.2.1 Maternal-fetal transfer by birth: Given the fact that Canadian women do not consume enough milk (15, 16), it is not surprising that over 1/3 of infants are born already deficient in vitamin D. In Manitoba, the PI has documented that 36% of infants from white or non-white parents are deficient in vitamin D at birth, defined as a serum 25(OH)D below 27.5 nmol/L, with 46% of their mothers themselves having values < 37.5 nmol/L (6). In that study, 20% of white infants were deficient, and as a group 60% of First Nations, Asian, Filipino and Black infants were deficient. This suggests that vitamin D deficiency is not uncommon, particularly in non-white women and their infants (6, 19-22). Likewise season of birth (19) and ethnicity (6) are important factors to consider in defining how much vitamin D is required to achieve and maintain target values for 25(OH)D in infants.

2.2.2 Infants from birth to 12 months: Infants have limited stores of vitamin D at birth because the amount transferred from the mother has a very short half life of 10-21 days (1). For infants exclusively breastfed, vitamin D supplementation is recommended by Health Canada (5) because vitamin D concentrations are low in the breast milk of Canadian mothers (4-40 IU/L). Fortified formula would provide ~ 400 IU vitamin D/L daily, but likely not achieved until close to 6 months of age (i.e., with intake 1L/d). After 6 months of age, the foods available to infants have limited vitamin D content.

2.3 Role of Early Life Vitamin D in Human Bone Health Term infants with 25(OH)D concentrations above 27.5 nmol/L have higher weight adjusted bone mass than those born with lower concentrations (6). The effects of higher maternal-fetal transfer of vitamin D are sustained long into childhood, as illustrated by a recent report from Southampton, UK (50N latitude): maternal vitamin D status in pregnancy, synonymous with fetal exposure to vitamin D in utero, was positively correlated with bone mass in the children measured as late as 9 years of age (3).

The effect of various dosages of vitamin D on whole body/skeletal bone mineral accretion in the first year of life has not been reported. In the first year of life, it is expected that whole body bone mineral content (BMC) will almost triple in parallel to growth (24, 25). In formula fed infants, whole body BMC at 1, 3, 6, 9 and 12 months of age are 79, 130, 160, 200 and 235 g respectively as measured with dual energy x-ray absorptiometry (DXA) with a precision error of 4.5% (25). Since the largest increment is between 1 and 3 months (63%), this is an ideal time to compare outcomes with respect to effects of various dosages of vitamin D on bone mineral accretion. However, this has yet to be conducted and is an important objective of the present proposal. It is anticipated that optimal vitamin D status will yield greater bone mass, since in Geneva, Switzerland (46N latitude), even a 400 IU/d vitamin D3 supplement in infancy (median duration of 12 months) is associated with higher BMD at 7 to 9 years of age (4). In the girls who received a vitamin D supplement in infancy, BMD was 6% higher in the distal radius and 9% higher in the femoral neck, even after adjustment for size (4). These positive associations must be viewed in conjunction with studies identifying peak bone mass as a critical factor in bone health (26). Whether the positive effects of the supplement translate into higher peak bone mass, is not yet known. An additional limitation is that no such studies have been conducted in Canada, with its unique climate, culture, food supply, and policies related to infant sun exposure. Since optimal vitamin D requirements for Canadian infants are ill defined, the benefits to bone mass are also unclear. As such, recommended dietary intake of vitamin D3 for Canadian infants must be identified by rigorous, well-controlled, randomized designs with optimal vitamin D status as the primary outcome.

2.4 New Paradigm for Optimal Vitamin D Status Physiologically, when blood calcium falls, PTH is released to promote hydroxylation of 25(OH)D to 1,25(OH)2D. Both PTH and 1,25(OH)2D mobilize of calcium (Ca) from bone and enhance absorption of Ca from the diet and glomerular filtrate. Elevated PTH levels characteristically seen in individuals with inadequate vitamin D status can result in the long latency disease of osteoporosis (27). A high PTH can also result from low dietary Ca, but for infants, breast milk and formula provide ample Ca.

Optimal 25(OH)D concentration for infants is unknown but is projected to be at least 75 nmol/L based on adult studies (8). This value is derived from well controlled dose-response studies of vitamin D3 supplementation in men and women, which demonstrate a reduction in serum PTH (8, 28, 29) with increasing 25(OH)D concentrations and a plateau in the mid-normal PTH reference range. However, current thinking suggests that the 25(OH)D-PTH dynamic is not the only instrument to determine recommendations, but should be supplemented with alternate biomarkers, such as bone mass and mineral metabolism, to more clearly define what is optimal (27). This is illustrated by a study of young adults in whom higher vitamin D concentrations (90-100 nmol/L) were associated with higher BMD when compared to those with lower concentrations (9). This would suggest that gains in 25(OH)D beyond those associated with the PTH plateau are important. Similarly, 25(OH)D concentration of 75 to 80 nmol/L in children 7 to 18 years of age are related to normalization of PTH (30-34) and has been selected as the target concentration for this age group as well. Concentrations of 25(OH)D at and above this value are associated with enhanced bone mineral accretion in one cohort (35) and in a randomized controlled trial (RCT) of vitamin D supplementation with 400 and 600 IU/d in adolescents (36). These studies again emphasize that the PTH-25(OH)D dynamic and bone mass are important determinants for establishing the RDA in pediatrics. Such dose-response studies of vitamin D3 do not exist for Canadian infants and it is possible that PTH should not be the only biomarker of adequacy during this life stage. There are limited dose-response studies [2] or RCT [1] examining daily oral vitamin D intake in infants (37-39). The details of these studies have recently been summarized as part of a NIH requested systematic review compiled by Canadian experts. The key message of this report is that there are no dose-response studies of vitamin D3 intake in infants, but only of vitamin D2 (9.5 x lower potency (12)) in dosages ranging from 100 to 1000 IU/d. These studies were of short duration and none were conducted in Canada. Additionally, not all studies measured PTH and none measured whole body bone mass. Clearly, a trial of vitamin D3 in Canadian infants is overdue.

In order to better understand how to optimize vitamin D status in infants, newer biomarkers of bone formation and resorption should be included to more comprehensively assess bone metabolism in association with 25(OH)D, PTH and whole body BMC. Suggested biomarkers include plasma osteocalcin and urinary N-telopeptide. Osteocalcin increases with growth and bone mineralization in the first year of life, as does alkaline phosphatase (40). Osteocalcin is the superior marker, since it also reflects seasonal changes in 25(OH)D and PTH in infancy (41). For bone resorption, urinary N-telopeptide is a practical marker, as it can be measured in urine and is also a specific index for bone resorption. Excretion of N-telopeptide in a spot urine sample in infants over the first year of life can be used with confidence for comparing groups of patients (42).

2.5 Safety Considerations, High Dosages Elevate 25(OH)D with No Adverse Effects There are no observed adverse effects at vitamin D2 or D3 doses of 1800 IU/d in infants (1). In the event of hypervitaminosis D, hypercalciuria and or hypercalcemia could occur. Sustained hypercalcemia could manifest as failure-to thrive, anorexia, irritability, nephrocalcinosis and its effects, and the remote possibility of cardiac arrhythmias. In one published study where infants received approximately 1200 IU of vitamin D per day (D2 supplements and D3 formula) (43), and in a pilot coordinated Dr. Taback (Univ. Manitoba) and the applicants (see CV module, CDA grant) where infants received 2000 IU/d of vitamin D3, no hypercalcemia or hypercalciuria was noted. In the later trial, PTH data are not yet available and this dose of vitamin D3 results in 25(OH)D well above 75 to 80 nmol/L (199 nmol/L, n=4). While too small to calculate SD, this study suggests that the required intake of vitamin D3 is likely below 2000 IU/D.

2.6 Theoretical Calculation of Vitamin D Intakes To Establish Study Dosage Groups As described in 2.1, the RDA is defined as the EAR + 2 SD and covers requirements of 97% of the population. If the target is 75 nmol/L for all infants, this means that the 2.5 percentile must be at this concentration. Using data from the PI's research of 83 cord blood samples, the mean value of 25(OH)D was 35 with SD of 15 nmol/L (full dataset from Weiler et al. (6)). Thus the lower 2.5 percentile is 5 nmol/L. To elevate this to 75 nmol/L, a gain in 70 nmol/L would be required (97 % of infants above target). Unfortunately, there is little available data as to the dose-response dynamics of mammalian cholecalciferol (D3) in infants, and studies of plant ergocalciferol (D2) may be misleading due to differences in bioavailability, which may be as much as a whole order of magnitude. The preliminary data from Drs. Taback and Weiler using daily supplements of either 400 IU or 2000 IU of D3 in a small number of Winnipeg infants (n=4 in each group) are the only data for us to base our estimates. Although too small a sample to confidently estimate measurement variance, they observed a rise of 44 and 115 nmol/L in the respective mean 25(OH)D concentrations in the first 3 months of supplementation. Thus, the 400 IU dose of vitamin D3 is expected to achieve a mean concentration of 75 nmol/L by 3 months of age. 800 IU D3 will be used in this study because this is currently recommended for Canadian infants. Because 2000 IU D3 was felt to be excessive based on the modest numbers of infants given this dose and their short follow up, we elected to select 1200 and 1600 IU as intermediate yet likely candidate RDA doses.

3.0 OBJECTIVES and HYPOTHESIS HYPOTHESIS: Daily oral dosage of 400 IU/d of vitamin D3 will be inadequate to achieve optimal vitamin D status in 97% of Canadian infants.

PRIMARY OBJECTIVE: To define the dosage of vitamin D3 required to achieve 25(OH)D concentrations ≥ 75 nmol/L at 3 months of age in exclusively breast fed infants.

SECONDARY OBJECTIVES: When multiple doses achieve our primary objective of optimal 25(OH)D concentrations, the best dosage will be identified based on: (i) 25(OH)D-PTH dynamics (ii) incidence of adverse events, such as disturbed mineral homeostasis (e.g. hypercalcemia, hypercalciuria, etc), and (iii) alternate markers of bone health (e.g. bone mass, osteocalcin and N-telopeptide) TERTIARY OBJECTIVE: We will examine the quantitative relationships between primary and secondary outcome measures and the various prospectively collected predictor variables, including dose, vitamin D from breast milk or fortified formulae, gender, season of birth, ethnicity, baseline vitamin D stores and determine if the selected dosage maintains 25(OH)D over the first year of life.

4.0 METHODOLOGY: Dose Response Study 4.1 Population n=192 breast-fed infants from greater Montreal region will be studied. The rationale for studying breast-fed infants is that this is the current recommended optimal food for infants, along with vitamin D supplements, and the fact that 85% of women in Canada initially breastfeed their infant (44, 45). Beginning with breastfeeding allows confirmation that the best dose is suitable while breastfeeding and if this dose is also optimal later in infancy with introduction of foods and weaning to vitamin D fortified formula. Initially a pilot study will be employed with 24 infants to evaluate the recruitment strategy, study questionnaires and procedures that will be used in the larger study.

4.2 Study Protocol 4.2.1 Recruitment: Rolling recruitment over 1 year with 1-year follow up for all beginning in September of 2006 and continuing through August 2007. Equal numbers across all months will be sought. At least two large pediatric clinics (Médicentre St-Lazare and Clinique de santé jeunesse) will be the primary recruitment centres with over 1500 newborns annually receive their ongoing medical care. These clinics provide care to families with a wide range of SES and cultures representative of Montreal and Canada. Infants will be recruited at the first postnatal visit at 2 weeks of age. Such recruitment age is suitable since breastfeeding will be deemed as established and recovery of birth weight and good health are confirmed. The clinician will inform women and families who meet inclusion criteria, and only those who are interested in participating in the study will have their names and contact address and telephone number forwarded to the study coordinator. All study visits will take place at the Mary Emily Clinical Nutrition Research Unit, School of Dietetics and Human Nutrition.

4.2.2 Study treatment groups: After obtaining written consent the infant will be randomized to a study group stratified for sex (see page 12) i for randomization process). At recruitment (2-4 weeks of age), baseline measurements will be conducted prior to providing treatment. Infants will then be randomized to receive 400, 800, 1200 or 1600 IU/d of vitamin D3 to 1 year of age. A placebo group is not included since the standard in Canada is 400 IU/d and a precedent for considering placebos unethical has already been set (37). The supplement will be double blinded to the investigators and all staff by coding of the supplements by Euro-Pharm who as agreed to provide the supplement in kind. This supplement will be stable for at least 3 months (the longest interval of measurements) and each dosage delivered in 2 ml volumes.

4.2.3 Frequency and duration of follow up: Baseline and all follow up visits (3, 6, 9, and 12 months of life) will include anthropometric measurements and blood and urine analysis for (25(OH)D, PTH, calcium, phosphorus, creatinine) as well as bone markers and bone mass measurements. An additional blood sample will be obtained 1 month after starting the study to monitor blood calcium levels. Bottles of the supplement will be assessed for compliance at these visits. Other sources of vitamin D intake will be reviewed by diet history as well as determining the content of vitamin D in the breast milk. Maternal baseline information regarding demographics will be gathered at the initial visit and dietary vitamin D intake will be assessed at each visit.

4.3 Details of Measurements INFANT: NUTRITIONAL AND HORMONAL STATUS AND BONE METABOLISM 4.3.1 Sample procurement: Blood and urine samples will be collected in infants at all visits. All samples will be taken between 8 and 10 am to control for diurnal variation permitting 3 to 4 infants to be seen in our Unit daily. Heparinized blood (~1 ml in infants via finger poke - 400 ul for safety, 600 ul for other measurements) and non-pharmacological approaches used to provide for pain control including swaddling and 1 ml 33% sucrose solution given sub lingual 2 minutes prior to collection (46).

4.3.2 25(OH)D and PTH concentrations: Vitamin D status will be measured using a RIA (25-50; Diasorin) that is known to measure both D2 and D3 in plasma (47). This method (RIA) is selected as the now most common clinical method over HPLC and competitive protein binding assays. Serum intact PTH will be measured using an ELISA (50 ul; Immutopics International).

4.3.3 Bone markers: Change in bone metabolism in response to 25(OH)D will be assessed by a marker of osteoblast activity related to mineralization, plasma osteocalcin (20 ul; Diasorin). Osteoclast activity will be assessed by measuring urinary N-telopeptide (ELISA, Osteomark) corrected to creatinine. The assay is specific to Type 1 collagen with a CV% <8%. N-telopeptide measurements urine selected over blood to reserve the small blood sample for other measurements. Urinary N-telopeptide in spot urine samples is a validated measurement in infancy (42). The PI is experienced in all of these measurements (6, 48).

4.3.4 Anthropometry: For infants, size at birth (weight, length, head circumference) and gestational age will be documented from the vaccine carnet. Growth will be assessed each visit using triplicate measurements of weight (to the nearest g without clothing/diaper), crown-heel length (to the nearest 0.1 cm using an infant length board) and head circumference (to the nearest 0.1 cm using a non-stretchable tape). Data will be expressed in absolute units and standard deviation scores using the data from the Centers for Disease Control at each age. Quality of growth achieved after term age will be available as lean and fat mass provided during measurement of bone mass using DXA, reported as accurate and reproducible (49).

4.3.5 Nutrition: Milk intake in infancy will be assessed by weighing infants prior to and after breast-feeding (i.e., test weighing and the basis of the required weigh scales). For this purpose, parents will be provided with electronic weigh scales designed for test weighing over 3 days then returned to the research site by courier. Additionally, breast milk vitamin D (all forms) will be measured (using HPLC (51, 52)) in samples collected at inception and the 3 month visit using an electronic breast pump. Mothers will be asked to feed the infant on one breast and pump from the other. Total intake of vitamin D will then be derived from milk intake and milk vitamin D concentration. Thus total intakes of vitamin D will be possible whether breast-fed or fed formula.

At each age, dietary and supplement intake will be documented in infants using written 3-day records that are designed to accommodate test weighing and documentation of other milks and any foods consumed as successfully used previously by the PI (53). Estimated portions sizes will be made using household measuring tools. Mothers will be asked about timing of introduction of solid foods or fluids other than breast-milk or vitamin D supplements. If infants wean to infant formula or cows milk, the product brand will be documented. It is anticipated that by 3 to 4 months of age that many infants will wean from breastfeeding to formula. However, the dosage will not be adjusted. Intake of vitamin D from infant formula, cows' milk etc will be documented and used to calculate total daily intake above the supplement. Such additional vitamin D will be addressed in the statistical analysis and is anticipated to be a systematic variation in total intakes.

4.3.6 Bone mass: Measurement of bone area, BMC and BMD of the whole body, lumbar vertebrae (L2-4) and femur at all visits will be conducted using DXA (QDR 4500A Discovery series, Hologic Inc.) at the Mary Emily Clinical Nutrition Research Unit. DXA has been validated for measuring infant whole body and regional BMC (49, 54, 55) and delivers minimal radiation (6 uSv) in comparison to standard pediatric x-rays (~60 uSv). Since positioning in infants is difficult to standardize, only BMC is used for whole body and femur. For lumbar spine, standardized positioning is feasible enabling assessment of bone area, BMC and BMD. Infants will not be sedated and will be scanned while sleeping and wrapped in a receiving blanket and standardized clothing without any metal zippers, clasps etc. Data will be expressed as absolute values for bone area, BMC and BMD and also as a rate of change for BMC. The measurement of whole body bone mass is ideal and recommended by ISCD (56). To enable complete data regarding bone, the next best measurement is lumbar spine, vertebra 1-4 (56). This measurement is easily attainable in infants to 1 year of age and only requires 30 to 60 seconds compared to whole body at 3 minutes. In addition, the femur can be scanned in 30 to 60 seconds and offers a novel assessment of a long bone. Whole body BMC will be corrected to body weight, length and lean mass and also expressed as change over the period of study. Correction to weight or length is endorsed by ISCD rather than more novel methods such as use of bone area and height (59) since normative data for infants is not currently available. Differences in whole body bone mineral accretion between inception, 3 and 6 months and between 6 and 12 months are greater than the error of measurement by DXA estimated at <4.5% (25, 49). Values for spine bone area, BMC and BMD and femur BMC will be compared among groups.

MATERNAL CHARACTERISTICS 4.3.7 General demographics and anthropometry include: Maternal age, weight gain in pregnancy, height, family income range and number of dependent members, employment, highest education level achieved, previous pregnancies, live births. To obtain accurate measurement of height, mothers will be measured at the inception visit. Weight will also be measured to accurately describe the population. Self-reported weight gain in pregnancy will be documented. Mothers will be asked to self-identify ethnicity. These data will be used to simply characterize the study population.

4.3.8 Nutrient intake: Dietary and supplement intake by the mothers during the last trimester of pregnancy will be assessed using a validated food frequency questionnaire, the modified Willett/Harvard (60). This questionnaire is modified to assess intakes over the last 3 months of pregnancy. These data will be used to describe vitamin D exposure of the fetus in utero when bone is mineralizing. At each visit and while the mother is lactating, intake of vitamin D will be assessed using a 24-hour recall. The value for maternal vitamin D intake will be used to describe our population as necessary to determine if results can be extrapolated to the Canadian population.

4.4 Recruitment and Statistical Analysis 4.4.1 Recruitment: Infants will be equally allocated to the 4 dosage groups, based on a randomization in blocks of 8 to accommodate stratifying by gender since growth diverges in male and female infants by the first year of life. Even distribution among the 4 seasons (standard calendar dates) will be sought by recruiting 1/12th of the sample each month. The fact that some infants may have already began vitamin D supplements will be considered as a systematic error.

4.4.2 Power and sample size: The sample size will be 48 to enable balanced groups across seasons and genders. This sample size will permit analysis of the data by feeding type: infants exclusively breast-fed versus weaning to formula as necessary to meet objective 3.

4.4.3 Data Analysis: The intention-to-treat principle will be applied, including all randomized infants for each outcome. For comparison purposes, results will also be evaluated in terms of the dose actually received. Should baseline imbalances occur between groups despite randomization, these will be treated as covariates and adjusted for. To compare proportions between treatment groups, sample proportions will be evaluated by a Chi-squared test of proportions, adjusted for multiple comparisons to ensure a family-wise error rate of 0.05. Results will be assessed at the each time point, with a Chi-squared test for trend in proportions to compare their temporal evolution. Mean 25(OH) D concentrations, bone mass, and biochemical indices of bone remodeling will be compared in each dose group under a fixed effects ANOVA model, with significant group differences localized by suitable post-hoc testing (e.g. Tukey method), again with adjustment for multiple comparisons to ensure a family-wise error rate of 0.05. Time course will be evaluated under a mixed effects ANOVA model (with the addition of time as a random effect). The dynamics of the 25(OH)D-PTH relationship is visually assessed in linearized log-log plots, whose slope is a measure of PTH sensitivity to 25(OH)D. The best-fit line is determined by least squares, and slopes compared by standard methods based on the distribution of regression coefficients as t-statistics. Taking the following as independent predictor variables - dose, source of vitamin D, age, gender, season of birth, ethnicity, and baseline vitamin D stores - their effect on the likelihood of achieving our therapeutic target will be evaluated by multiple logistic regression, with ordinary multivariate linear regression to examine their impact on serum concentration of 25(OH)D, bone mass, osteocalcin, and N-telopeptide.

ELIGIBILITY:
Inclusion Criteria:

* Healthy singleton term born infants of appropriate size for gestational age (AGA) according to the Centers for Disease Control growth charts based on weight at birth between the 5th and 95th percentiles for sex; and born to healthy breastfeeding women. This allows us to assess growth and bone mineral accretion without bias of intrauterine growth restriction.

Exclusion Criteria:

* Infants of mothers with history of gestational diabetes or hypertension in pregnancy; chronic alcohol use; malabsorption syndromes due to malabsorption of vitamin D (celiac disease, Crohn's etc.); and multiple births.
* Should any exclusion criteria be identified after recruitment, the infant will be excluded from the main analyzes, but followed in a separate arm as intent-to-treat.

Ages: 2 Weeks to 5 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 132 (Actual)
Dates: Start 2007-03; Primary Completion 2011-09 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Vitamin D plasma concentrations | 12 months
  25(OH)D concentrations will me measured in infants over the first year of life. The blood sampling will be done at 1, 2, 3, 6, 9 and 12 months of age. Monitoring the vitamin D concentrations will allow the investigators to determine the best dose of vitamin D for breast fed infants receiving one of three vitamin D dosages.

SECONDARY OUTCOMES:
Bone mineral content | 12 months
  Bone mineral content will be assessed at 1, 3, 6, 9 and 12 months of age. Using DXA technology which provides measures of bone mineral content as well as body composition measurements the investigators will be able to correlate these changes with vitamin D concentrations.

CONTACTS AND LOCATIONS:
Overall Officials: Hope A Weiler, PhD, Principal Investigator — McGill University; Celia Rodd, MD, Principal Investigator — Montreal Children's Hospital of the MUHC
Locations (1):
- Mary Emily Clinical Nutrition Research Unit, Sainte-Anne-de-Bellevue, Quebec, Canada

REFERENCES:
- [Derived] Gharibeh N, Gallo S, Sotunde OF, Vanstone CA, Rodd CJ, Weiler HA. Patterns of Bone Mineral Accretion and Sex Differences in Healthy Term Vitamin D Replete and Breastfed Infants From Montreal, Canada: Bone Mass Reference Data. J Clin Densitom. 2022 Jan-Mar;25(1):43-53. doi: 10.1016/j.jocd.2021.07.004. Epub 2021 Jul 24. PMID 34479797
- [Derived] Huey SL, Acharya N, Silver A, Sheni R, Yu EA, Pena-Rosas JP, Mehta S. Effects of oral vitamin D supplementation on linear growth and other health outcomes among children under five years of age. Cochrane Database Syst Rev. 2020 Dec 8;12(12):CD012875. doi: 10.1002/14651858.CD012875.pub2. PMID 33305842
- [Derived] Mok E, Vanstone CA, Gallo S, Li P, Constantin E, Weiler HA. Diet diversity, growth and adiposity in healthy breastfed infants fed homemade complementary foods. Int J Obes (Lond). 2017 May;41(5):776-782. doi: 10.1038/ijo.2017.37. Epub 2017 Feb 6. PMID 28163319
- [Derived] Hazell TJ, Gallo S, Berzina I, Vanstone CA, Rodd C, Weiler HA. Plasma 25-hydroxyvitamin D, more so than its epimer, has a linear relationship to leaner body composition across infancy in healthy term infants. Appl Physiol Nutr Metab. 2014 Oct;39(10):1137-43. doi: 10.1139/apnm-2013-0586. Epub 2014 May 1. PMID 25004404
- [Derived] Gallo S, Comeau K, Vanstone C, Agellon S, Sharma A, Jones G, L'Abbe M, Khamessan A, Rodd C, Weiler H. Effect of different dosages of oral vitamin D supplementation on vitamin D status in healthy, breastfed infants: a randomized trial. JAMA. 2013 May 1;309(17):1785-92. doi: 10.1001/jama.2013.3404. PMID 23632722